CLINICAL TRIAL: NCT05310292
Title: A Glucometabolic Evaluation of Patients With Idiopathic Ketotic Hypoglycemia
Acronym: IKH_MetEx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Frederik Gluud Grøndahl, Principal investigator, Medical Doctor, PhD student, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-21056987
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Idiopathic Ketotic Hypoglycemia
Keywords: Idiopathic ketotic hypoglycemia; Glucose metabolism; Gut homones; Amino acids; Glucagon; Insulin; Continuous glucose monitor; CGM; Oral glucose tolerance test; Mixed meal test
MeSH Terms: conditions — Insulin Resistance | interventions — Glucose Tolerance Test; 2-methylcyclopentadienyl manganese tricarbonyl

STUDY DESIGN:
Intervention Model Description: A case-control intervention study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects diagnosed with IKH (Experimental): 10 patients, diagnosed with IKH
  Interventions: Biological: Oral glucose tolerance test; Biological: Mixed meal test
- Healthy control subjects (Experimental): 10 subjects, healthy, matched for gender, BMI, age
  Interventions: Biological: Oral glucose tolerance test; Biological: Mixed meal test

INTERVENTIONS:
Biological: Oral glucose tolerance test — Consumption of 75 grams of glucose, diluted in water, added 1,5 g of acetaminophen.
  Other Names: OGTT
Biological: Mixed meal test — Consumption of a standardized liquid meal, with caloric and dietary content equal to a standard meal.
  Other Names: MMT

SUMMARY:
The project will evaluate 1) the postprandial metabolism and 2) continuous glucose levels in subjects diagnosed with Idiopathic Ketotic Hypoglycemia (IKH)) and healthy control subjects.

DETAILED DESCRIPTION:
IKH is a common, but not fully understood, condition in children, and in some the condition may persist in adulthood. In the present study we seek to evaluate the postprandial metabolism in adult subjects diagnosed with IKH through a clinical study including:

1. two test days, where the subjects completes a) an oral glucose tolerance test (OGTT) and b) a miced meal test (MMT). Before, during and after ingestion of the OGTT/MMT, blood samples will be frequently drawn for the evaluation of plasma glucose, hormones, amino acids and more. During both tests, the subjects will recieve a continuous infusion of primed glucose tracer to further evaluate the glucose metabolism.
2. a 14-day period where the subjects will lead the usual lives, wearing a continuous glucose monitor (CGM). This will enable us to evaluate long-term differences in plasma glucose levels in IKH.

ELIGIBILITY:
Inclusion Criteria:

* IKH-participants:
* Verified diagnosis of IKH by health professional
* BMI of 18-30 kg/m2
* Normal liver- and kidney function
* informed consent

Healthy control participants

* Normal glucose tolerance
* BMI of 18-30 kg/m2
* Normal liver- and kidney function
* informed consent

Exclusion Criteria:

* A history of diabetes
* close family members with diabetes
* use of drugs affecting the glucose metabolism that cannot be paused
* anemia
* any condition that the study investigators deem unacceptable for participation
* pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose | -120, -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
  The intergroup difference in peak to nadir difference in plasma glucose following OGTT/MMT
Time in range (CGM) | 0-14 days of CGM-period
  The intergroup difference in time spend in glycemic range, measured by CGM

SECONDARY OUTCOMES:
Endogenous glucose production | -120,, -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
  Rate of appearance of glucose, measured by tracer dilution technique
Glucose revomal | -120, -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
  Rate of disappearance of glucose, measured by tracer dilution technique
Amino acids | -120,-60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
  Plasma concentrations of amino acids
Insulin | -120,-60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
  Plasma concentrations of insulin
Glucagon | -120,-60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
  Plasma concentrations of glucagon
Glucagon like peptide-1 (GLP-1) | -120,-60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
  Plasma concentrations of GLP-1
Glucose-dependent insulinotropic polypeptide (GIP) | -120,-60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes
  Plasma concentrations of GIP
Coefficients of variation (CV) of plasma glucose | 0-14 days of CGM-period
  CV of plasma glucose measured by CGM
Mean plasma glucose | 0-14 days of CGM-period
  Average value of plasma glucose measured by CGM
Risk of hypoglycemia | 0-14 days of CGM-period
  Time spend in hypoglycemia measured by CGM

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Department of Medicine, Gentofte Hospital, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No